CLINICAL TRIAL: NCT03014063
Title: Vasopressin Plasma Concentrations in Responders and Non-responders to Exogenous Vasopressin Infusion in Patients With Septic Shock
Brief Title: Vasopressin Plasma Concentrations in Patients Receiving Exogenous Vasopressin Infusion for Septic Shock
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1254
Record Dates: First submitted 2017-01-04; First posted 2017-01-09 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Septic Shock
Keywords: sepsis; septic shock; vasopressin; AVP
MeSH Terms: conditions — Shock, Septic; Sepsis; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma vasopressin concentration in patients receiving exogenous vasopressin
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemodynamic responders: Those with a mean arterial pressure of at least 65mmHg and a decrease in catecholamine dose (in norepinephrine equivalents) from initiation of exogenous vasopressin therapy to the time of the sample collection used for analysis of plasma vasopressin concentration
- Hemodynamic non-responders: Those without a mean arterial pressure of at least 65mmHg and/or a decrease in catecholamine dose (in norepinephrine equivalents) from initiation of exogenous vasopressin therapy to the time of the sample collection used for analysis of plasma vasopressin concentration

SUMMARY:
This is a prospective observational cohort trial evaluating a single plasma vasopressin concentration in patients receiving exogenous, adjunctive vasopressin for septic shock. The trial is designed to determine whether plasma vasopressin concentration influences the likelihood of hemodynamic response to exogenous vasopressin therapy.

DETAILED DESCRIPTION:
Vasopressin is an endogenous hormone that decreases serum osmolarity and increases blood pressure. As a part of the stress response to hypotension, vasopressin is released from the posterior pituitary and leads to vasoconstriction through agonism of the vascular vasopressin V1 receptor. In patients with septic shock, endogenous vasopressin levels are initially elevated but quickly fall to levels at or below those of normal physiology (1.4-3.6pg/mL) because of the depletion of endogenous store. Sharshar et al. evaluated two sets of patients with septic shock, one of which was evaluated earlier in the septic shock course (3.6 ± 2.3 hours, n=18) and one evaluated at a later time from shock onset (mean 38.7 ± 28.4 hours, n=44). The group of patients evaluated earlier in their septic shock course were more likely than patients evaluated later to have elevated (>3.6 pg/mL) plasma vasopressin levels (88.9% vs. 38.6%, respectively). Similarly, a case series evaluated single vasopressin levels in three patients with septic shock, one of whom was in the first day of shock onset and two of whom were in the fifth and sixth day of shock onset. The patient in the earlier stages of septic shock had a plasma vasopressin level that was increased (16pg/mL), while the two patients in the later stages of septic shock had decreased plasma vasopressin levels (1.6 and 1.8pg/mL). The exact timing of when patients transition from having elevated endogenous vasopressin levels to having normal levels of vasopressin is currently unclear. In a clinical trial enrolling patients within the first 12 hours of shock onset, median endogenous vasopressin levels were 3.5 pg/mL (interquartile range 1.8, 5.3 pg/mL; n=54). Some have even hypothesized that vasopressin levels rise before clinical hypotension is apparent and the decline in vasopressin levels is associated with the onset of apparent hypotension. Further complicating this issue, endogenous vasopressin levels have been shown to be lower in patients with septic shock compared to other shock etiologies such cardiogenic shock (3.1 ± 1pg/mL in patients with septic shock vs. 22.7 ± 2.2pg/mL in patients with cardiogenic shock, p<0.001). The etiology of this discrepancy in endogenous vasopressin response by shock type is unclear, but a "relative deficiency" of vasopressin is theorized to exist in patients with septic shock.

In light of these findings, exogenous arginine vasopressin (AVP) has been added to exogenous catecholamines to increase mean arterial pressure (MAP) and to decrease catecholamine requirements in patients with vasodilatory shock. The use of AVP for these purposes in patients with septic shock is in keeping with the Surviving Sepsis Campaign Guidelines. In the Vasopressin and Septic Shock Trial (VASST), low-dose AVP was infused at a rate of 0.01-0.03 units/min in combination with norepinephrine to achieve a goal MAP of 65-75mmHg. Plasma vasopressin levels in patients receiving AVP were elevated at 6 (68.3pg/mL) and 24 hours (90.5pg/mL) in comparison to patients not receiving AVP (3.0pg/mL at baseline with no significant change at 6 or 24 hours). Association of plasma vasopressin levels with hemodynamic response to AVP, though, was not evaluated in VASST.

Concomitant corticosteroid use has been observed to decrease the total dose of administered AVP, to increase the proportion of patients alive and free of vasopressors at day 7, to increase plasma vasopressin concentrations by 33% at 6 hours and 67% at 24 hours, and to lead to lower 28- and 90-day mortality (35.9% vs. 44.7%, p=0.03 and 42.5% vs. 55.5%, p=0.01, respectively) than in those that received AVP alone. These findings generated the hypothesis that concomitant administration of AVP and corticosteroids results in increased plasma vasopressin levels versus AVP administration alone, leading to positive clinical outcomes in septic shock. Furthering the hypothesis that plasma vasopressin levels may influence outcomes in septic shock, genetic differences in leucyl/cystinyl aminopeptidase, the primary vasopressin metabolic enzyme, have been associated with more rapid vasopressin clearance, lower plasma vasopressin levels, and increased mortality in patients with septic shock. However, a study evaluating vasopressin plasma concentrations in patients with multiple shock types not administered exogenous AVP observed higher vasopressin concentrations in those with hemodynamic dysfunction than in those without (mean 14.1 ± 26 vs. 8.7 ± 10.8pg/mL, respectively) regardless of shock type. This suggests that plasma vasopressin concentration may not directly correlate with MAP.

The impact of body mass (which may influence vasopressin levels when fixed-dose AVP is administered) on hemodynamic response to AVP has been inconsistent. Studies have observed a negative correlation between BMI and change in MAP at 6 hours and a correlation between increasing weight-adjusted AVP dose and reduction in catecholamine requirements, suggesting that hemodynamic response to AVP is associated with body mass. In contrast, a third study observed no association between BMI and AVP dose required to meet goal MAP when AVP was administered as the sole vasopressor. Finally, a fourth found an inverse correlation between BMI and APACHE II-adjusted 28-day mortality, regardless of the fact that overweight and obese patients received less weight-adjusted vasopressin than underweight or normal weight patients. This suggests that while BMI may impact plasma vasopressin concentration, the change in vasopressin concentration may not have an impact on clinical outcomes.

Recently, a retrospective study was completed at the Cleveland Clinic to evaluate predictors of hemodynamic response to fixed-dose AVP in patients with septic shock. Patients were considered to be responders to AVP if a decrease in catecholamine dose was achieved with MAP≥65mmHg at 6 hours. The overall response rate to fixed-dose vasopressin was 45.4%. Within this study, only admission to surgical or neurosciences intensive care units (ICU) vs. medical ICU and lower lactate level were associated with increasing chance of response to AVP (OR 1.71, 95% CI 1.175-2.463, p=0.0049 and OR 0.925, 95% CI 0.887-0.965, p=0.0003, respectively) on logistic regression. Factors previously found to impact vasopressin levels (such as concomitant use of corticosteroids) were not associated with hemodynamic response. However, plasma vasopressin levels were not evaluated in this retrospective study.

The relationship between plasma vasopressin concentration and hemodynamic response in patients receiving AVP is unclear. While concomitant corticosteroids have been observed to increase plasma vasopressin concentrations, corticosteroids themselves have been shown to shorten time in septic shock, possibly confounding any relationship between plasma vasopressin concentration and hemodynamic response in patients receiving both agents. As previously mentioned, data correlating body mass with hemodynamic response have been inconsistent, but vasopressin levels in patients receiving fixed dose AVP seem to be lower in patients with higher body mass. The recent study at the Cleveland Clinic found no association between factors associated with increased plasma vasopressin level and hemodynamic response. Together, these data call into question the idea of a dose-response relationship between plasma vasopressin concentration and hemodynamic response. This study seeks to prospectively evaluate whether plasma vasopressin levels are associated with improved rates of hemodynamic response to fixed-dose AVP therapy in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Patients with septic shock as defined by The Third International Consensus Definitions for Sepsis and Septic Shock
* Patients ≥18 years of age
* Treatment with exogenous vasopressin, as ordered by the primary medical team, at a constant infusion rate for at least 3 hours as an adjunctive vasopressor to catecholamine therapy
* Admission to a medical, surgical, or neurosciences intensive care unit
* Presence of a central venous catheter or arterial line (as determined by the primary medical team)

Exclusion Criteria:

* Patients treated with vasopressin for indications other than septic shock
* Patients administered vasopressin that is titrated within the first 3 hours
* Patients receiving vasopressin as the sole vasoactive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with septic shock that are receiving fixed-dose exogenous vasopressin as an adjunct to catecholamines
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Plasma vasopressin concentration | 3-6 hours from initiation of exogenous vasopressin administration

SECONDARY OUTCOMES:
Mean arterial pressure | Analyzed at time of vasopressin blood draw, 3-6 hours from initiation of exogenous vasopressin administration
Catecholamine dose in norepinephrine equivalents | Analyzed at time of vasopressin blood draw, 3-6 hours from initiation of exogenous vasopressin administration
ICU mortality | Analyzed at ICU discharge, up to 1 year
In-hospital mortality | Analyzed at hospital discharge, up to 1 year
Vasopressor-free days | Day 14
ICU-free days | Day 14
Acute kidney injury | Analyzed at ICU discharge, up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Russell JA. Bench-to-bedside review: Vasopressin in the management of septic shock. Crit Care. 2011 Aug 11;15(4):226. doi: 10.1186/cc8224. PMID 21892977
- [Background] Sharshar T, Blanchard A, Paillard M, Raphael JC, Gajdos P, Annane D. Circulating vasopressin levels in septic shock. Crit Care Med. 2003 Jun;31(6):1752-8. doi: 10.1097/01.CCM.0000063046.82359.4A. PMID 12794416
- [Background] Sharshar T, Carlier R, Blanchard A, Feydy A, Gray F, Paillard M, Raphael JC, Gajdos P, Annane D. Depletion of neurohypophyseal content of vasopressin in septic shock. Crit Care Med. 2002 Mar;30(3):497-500. doi: 10.1097/00003246-200203000-00001. PMID 11990905
- [Background] Bauer SR, Lam SW. Arginine vasopressin for the treatment of septic shock in adults. Pharmacotherapy. 2010 Oct;30(10):1057-71. doi: 10.1592/phco.30.10.1057. PMID 20874043
- [Background] Russell JA, Walley KR, Singer J, Gordon AC, Hebert PC, Cooper DJ, Holmes CL, Mehta S, Granton JT, Storms MM, Cook DJ, Presneill JJ, Ayers D; VASST Investigators. Vasopressin versus norepinephrine infusion in patients with septic shock. N Engl J Med. 2008 Feb 28;358(9):877-87. doi: 10.1056/NEJMoa067373. PMID 18305265
- [Background] Lin IY, Ma HP, Lin AC, Chong CF, Lin CM, Wang TL. Low plasma vasopressin/norepinephrine ratio predicts septic shock. Am J Emerg Med. 2005 Oct;23(6):718-24. doi: 10.1016/j.ajem.2005.02.055. PMID 16182977
- [Background] Landry DW, Levin HR, Gallant EM, Ashton RC Jr, Seo S, D'Alessandro D, Oz MC, Oliver JA. Vasopressin deficiency contributes to the vasodilation of septic shock. Circulation. 1997 Mar 4;95(5):1122-5. doi: 10.1161/01.cir.95.5.1122. PMID 9054839
- [Background] Tsuneyoshi I, Yamada H, Kakihana Y, Nakamura M, Nakano Y, Boyle WA 3rd. Hemodynamic and metabolic effects of low-dose vasopressin infusions in vasodilatory septic shock. Crit Care Med. 2001 Mar;29(3):487-93. doi: 10.1097/00003246-200103000-00004. PMID 11373409
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Background] Gordon AC, Mason AJ, Perkins GD, Stotz M, Terblanche M, Ashby D, Brett SJ. The interaction of vasopressin and corticosteroids in septic shock: a pilot randomized controlled trial. Crit Care Med. 2014 Jun;42(6):1325-33. doi: 10.1097/CCM.0000000000000212. PMID 24557425
- [Background] Southard RE, Boyle WA. Corticosteroids and the original vasopressin and septic shock trial subgroups. Crit Care Med. 2010 Jan;38(1):338; authore reply 338-9. doi: 10.1097/CCM.0b013e3181bc7ab8. No abstract available. PMID 20023496
- [Background] Bauer SR, Lam SW, Cha SS, Oyen LJ. Effect of corticosteroids on arginine vasopressin-containing vasopressor therapy for septic shock: a case control study. J Crit Care. 2008 Dec;23(4):500-6. doi: 10.1016/j.jcrc.2008.04.002. Epub 2008 Jun 30. PMID 19056013
- [Background] Russell JA, Walley KR, Gordon AC, Cooper DJ, Hebert PC, Singer J, Holmes CL, Mehta S, Granton JT, Storms MM, Cook DJ, Presneill JJ; Dieter Ayers for the Vasopressin and Septic Shock Trial Investigators. Interaction of vasopressin infusion, corticosteroid treatment, and mortality of septic shock. Crit Care Med. 2009 Mar;37(3):811-8. doi: 10.1097/CCM.0b013e3181961ace. PMID 19237882
- [Background] Torgersen C, Luckner G, Schroder DC, Schmittinger CA, Rex C, Ulmer H, Dunser MW. Concomitant arginine-vasopressin and hydrocortisone therapy in severe septic shock: association with mortality. Intensive Care Med. 2011 Sep;37(9):1432-7. doi: 10.1007/s00134-011-2312-3. Epub 2011 Jul 21. PMID 21779849
- [Background] Nakada TA, Russell JA, Wellman H, Boyd JH, Nakada E, Thain KR, Thair SA, Hirasawa H, Oda S, Walley KR. Leucyl/cystinyl aminopeptidase gene variants in septic shock. Chest. 2011 May;139(5):1042-1049. doi: 10.1378/chest.10-2517. Epub 2011 Feb 17. PMID 21330387
- [Background] Jochberger S, Mayr VD, Luckner G, Wenzel V, Ulmer H, Schmid S, Knotzer H, Pajk W, Hasibeder W, Friesenecker B, Mayr AJ, Dunser MW. Serum vasopressin concentrations in critically ill patients. Crit Care Med. 2006 Feb;34(2):293-9. doi: 10.1097/01.ccm.0000198528.56397.4f. PMID 16424705
- [Background] Miller JT, Welage LS, Kraft MD, Alaniz C. Does body weight impact the efficacy of vasopressin therapy in the management of septic shock? J Crit Care. 2012 Jun;27(3):289-93. doi: 10.1016/j.jcrc.2011.06.018. Epub 2011 Aug 19. PMID 21855282
- [Background] Hodge EK, Hughes DW, Attridge RL. Effect of Body Weight on Hemodynamic Response in Patients Receiving Fixed-Dose Vasopressin for Septic Shock. Ann Pharmacother. 2016 Oct;50(10):816-23. doi: 10.1177/1060028016656384. Epub 2016 Jun 23. PMID 27340145
- [Background] Lam SW, Bauer SR, Cha SS, Oyen LJ. Lack of an effect of body mass on the hemodynamic response to arginine vasopressin during septic shock. Pharmacotherapy. 2008 May;28(5):591-9. doi: 10.1592/phco.28.5.591. PMID 18447658
- [Background] Wacharasint P, Boyd JH, Russell JA, Walley KR. One size does not fit all in severe infection: obesity alters outcome, susceptibility, treatment, and inflammatory response. Crit Care. 2013 Jun 20;17(3):R122. doi: 10.1186/cc12794. PMID 23786836
- [Background] Annane D, Sebille V, Charpentier C, Bollaert PE, Francois B, Korach JM, Capellier G, Cohen Y, Azoulay E, Troche G, Chaumet-Riffaud P, Bellissant E. Effect of treatment with low doses of hydrocortisone and fludrocortisone on mortality in patients with septic shock. JAMA. 2002 Aug 21;288(7):862-71. doi: 10.1001/jama.288.7.862. PMID 12186604
- [Background] Sprung CL, Annane D, Keh D, Moreno R, Singer M, Freivogel K, Weiss YG, Benbenishty J, Kalenka A, Forst H, Laterre PF, Reinhart K, Cuthbertson BH, Payen D, Briegel J; CORTICUS Study Group. Hydrocortisone therapy for patients with septic shock. N Engl J Med. 2008 Jan 10;358(2):111-24. doi: 10.1056/NEJMoa071366. PMID 18184957
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Sacha GL, Lam SW, Duggal A, Torbic H, Bass SN, Welch SC, Butler RS, Bauer SR. Predictors of response to fixed-dose vasopressin in adult patients with septic shock. Ann Intensive Care. 2018 Mar 6;8(1):35. doi: 10.1186/s13613-018-0379-5. PMID 29511951